CLINICAL TRIAL: NCT07274254
Title: Lidocaine for Opioid Sparing in Vaso-occlusive Crisis of Sickle Cell Disease
Acronym: LidoVOC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC24_0427
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Vaso-Occlusive Pain Episode in Sickle Cell Disease
Keywords: Sickle Cell disease; Sickle Cell Syndrome; Vaso-occlusive crisis; Acute Chest Syndrome; Painful crisis; Pain management; Opioid sparing; Lidocaine
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome; Agnosia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Controlled, radomized, Double blinded, Prospective, Superiority
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Lidocaine + standard of care (Experimental): Lidocaine hydrochloride 20 mg/mL, solution, 20 mL ampoule for intravenous administration Administration : parenteral route on peripheral or central venous catheter.
  * Bolus of 1.5 mg/kg bolus during 30 minutes, with a maximum dose of 180 mg (18mL)
  * Immediately followed by a continuous infusion of 1 mg/kg/h (max 120mg/h =- 12mL/h) during 72 hours.
  Interventions: Drug: Lidocain; Drug: Standard of care
- Control group: placebo + standard of care (Placebo Comparator): Placebo is 20 mL ampoules of sodium chloride (NaCl 0.9%) for injection. Administration : parenteral route on peripheral or central venous catheter.
  * Bolus of 1.5 mg/kg bolus during 30 minutes, with a maxium dose of 180 mg (18mL)
  * Immediately followed by a continuous infusion of 1 mg/kg/h (max 120mg/h = 12mL/h) during 72 hours.
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Lidocain — Lidocaine hydrochloride 20 mg/mL, solution, 20 mL ampoule for IV administration (25 ampoules) Administration : parenteral route on peripheral or central venous catheter. - Bolus of 1.5 mg/kg bolus dur
  Arms: Experimental group: Lidocaine + standard of care
Drug: Placebo — Placebo is 20 mL ampoules of sodium chloride (NaCl 0.9%) for injection Administration : parenteral route on peripheral or central venous catheter.
  * Bolus of 1.5 mg/kg bolus during 30 minutes, with a maxium dose of 180 mg (18mL)
  * Immediately followed by a continuous infusion of 1 mg/kg/h (max 120mg/h = 12mL/h) during 72 hours.
  Arms: Control group: placebo + standard of care
Drug: Standard of care — Standard of care

SUMMARY:
The purpose of the study is to determine whether adding lidocaine to standard of care in pain management during severe vaso-occlusive crisis has an effect on the cumulative opioid consumption expressed as morphine milligram equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Known sickle cell disease with an SS, SC, Sβ, or Sβ+ genotype
* Patient admitted to the Intensive Care Unit for Vaso-Occlusive Crisis and/or ACS as the main reason for admission:

  * Vaso-Occlusive Crisis defined by acute pain or tenderness, affecting at least one part of the body, including limbs, ribs, sternum, head (skull), spine, and/or pelvis, not attributable to other causes
  * Acute Chest Syndrome defined by the association of clinical respiratory sign(s): dyspnea and/or chest pain and/or auscultatory abnormality (crepitants and/or bronchial breathing) with a new pulmonary infiltrate on chest X-ray, thoracic CT-scan, or lung ultrasound.
* Treatment with parenteral morphine or oxycodone started less than 72 hours prior to inclusion
* Patient or next of kin informed about the study and having consented to the participation of the patient in the study. If patient is no competent and no next of kin can be contacted during screening for the study, trial inclusion will be completed as an emergency procedure by the Intensive Care Unit physician, in compliance with French law.
* French speaking
* Patient with health care insurance

Exclusion Criteria:

* Pregnant women or nursing mothers; Women of child bearing potential will be tested for pregnancy before inclusion
* Patients under guardianship, curatorship or under legal protection
* Prisoners or subjects who are involuntarily incarcerated
* Sickle Cell Disease acute complication other than Vaso-Occlusive Crisis or Acute Chest Syndrome as the main reason for admission:

priapism, stroke, acute splenic sequestration, acute hepatic sequestration, bone marrow necrosis…

* Patients wearing a lidocaine-medicated plaster at the time of screening for inclusion
* Known or assumed hypersensitivity to lidocaine hydrochloride, other local anaesthetics (e.g., bupivacaine or ropivacaine) or an excipient
* Patients treated with anti-arhythmic drugs known to induce torsade de pointe.
* Patients on chronic or occasional treatment with drugs that interact with the 3A cytochrome isoenzymes (CYP3A) and/or 1A2 cytochrome isoenzymes (CYP1A2)
* Patients with recurrent porphyria, porphyria in remission, or known asymptomatic carriage of gene mutations responsible for porphyria
* Epileptic patients
* Hypovolemic shock or shock of other cause at screening for inclusion
* Known atrioventricular block, QT prolongation or other heart conduction disorder or heart failure
* Chronic respiratory failure with long term non invasive ventilation (excluding Continuous Positive Air way pressure), or long term oxygen therapy at home
* Acute Respiratory Distress Syndrome according to The 2012 Berlin definition
* Acute or Chronic liver failure with MELD > 19 according to CKD-EPI
* Acute or Chronic kidney failure with clearance <30mL/min/m2
* Body weight <40kg and >120kg
* Prior inclusion in the study in the last 3 months
* Patient under invasive mechanical ventilation
* Altered consciousness with Glasgow coma scale <13

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative parenteral opioid dose between randomization and discharge from the intensive care unit expressed in morphine milligram equivalent. | up to 28 days
  To determine whether adding lidocaine to the standard of care in pain during severe vaso-occlusive crisis has an effect on the cumulative opioid consumption expressed as morphine milligram equivalent (MME)

SECONDARY OUTCOMES:
Intensive Care Unit length of stay | up to 28 days
hospital length of stay | up to 28 days
Visual analogue pain Scale score during Intensive Care Unit stay | up to 28 days
  Compare between groups the pain intensity as evaluated using a Visual Analogue pain Scale from 0 (no pain) to 10 (very intense pain).
Categorical Pain Score during Intensive Care Unit stay | up to 28 days
  Compare between groups the pain intensity as evaluated using Categorical Pain Score (CPS)
Time of resolution of severe vaso-occlusive crisis | up to 28 days
  presence of at least three of the following four criteria:
  * continuous apyrexia for the last 8 hours,
  * no need for intravenous opioid infusion for the last 8 hours,
  * ability to walk or move without pain,
  * absence of spontaneous pain with a CPS ≤1
time to last parenteral opioid dose | up to 28 days
  Time from randomisation to the last parenteral opioid dose
vaso-occlusive crisis complications during Intensive Care Unit stay | up to 28 days
  secondary acute chest syndrome
vaso-occlusive crisis complications during Intensive Care Unit stay | up to 28 days
  need for blood transfusion
vaso-occlusive crisis complications during Intensive Care Unit stay | up to 28 days
  need for red blood cell exchange
vaso-occlusive crisis complications during Intensive Care Unit stay | up to 28 days
  need for life-supporting therapies defined as invasive mechanical ventilation or dialysis or vasopressor support
quality of life with reduced impact of Sickle Cell Disease on health | At Day 28
  Score of French version of Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me).
  It is a patient-reported outcome measurement system with a 39 items questionnaire, assessing several aspects of SCD impact on general health state. For the present study, the questionnaires regarding emotional impact, pain episodes, pain impact, Social Functionning will be used.
safety profile of lidocaine infusion | at 28 days
  Compare between groups safety profile of lidocaine infusion at D28
Rate of readmission for vaso-occlusive crisis after Intensive Care Unit discharge | At day 28
  Frequency of any adverse events and frequency of serious adverse events
Assess the economic efficiency of lidocaine added to standard of care compared to standard of care alone | At day 28
  Incremental cost-effectiveness ratio (cost per Quality-Adjusted Life-Year, QALY) comparing lidocaine + standard of care (SOC) to SOC alone

CONTACTS AND LOCATIONS:
Locations (11):
- France (10):
  - CHU Bordeaux, Bordeaux
  - CHU Lille, Lille
  - CHU La Timone, Marseille
  - CHU de Nantes, Nantes
  - CHU Orléans, Orléans
  - Hôpital Tenon APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen, Rouen
  - Oncopole Toulouse, Toulouse
  - CHRU Tours - Hôpital Bretonneau, Tours
- CHU Guadeloupe, Les Abymes, Guadeloupe